CLINICAL TRIAL: NCT03901781
Title: A Dose-escalating Phase 1 Open-label Safety Study of ST266 Given by Non-invasive Intranasal Trans-cribriform Delivery in Glaucoma Suspect Subjects Without Evidence of Glaucomatous Damage.
Brief Title: Study of ST266 Given by Intranasal Delivery in Glaucoma Suspect Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST266-IOPHTN-101
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: This clinical trial is a dose escalating design in three (3) cohorts of three (3) subjects per Cohort. In the first cohort, subjects will be administered ST266, delivered intranasally, at a dose of two hundred microliters (200 µL) daily for 14 days, in alternating single nostrils. After 14 daily treatments there is a seven (7)-day follow-up period. If there are no SAEs and no pattern of concern in the AE's, the Investigator may proceed to the second cohort of three (3) subjects. In Cohort Two, three (3) subjects will be administered 200 µL to each nostril daily (400 µL total per day) for 14 days. There will be a seven (7)-day follow-up. Like Cohort One, if there are no safety concerns, the investigator may move on to the third cohort of three (3) subjects. In Cohort Three, three (3) subjects will be administered 200 µL to each nostril daily (400 µL total per day) for 28 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Cohort One (Experimental): Three (3) subjects, ST266 200 µL administered by trans-cribriform intranasal device once a day for 14 days using alternating sides (nostrils) with a follow-up visit at seven (7) days following End of Treatment (EOT), a follow-up call at one (1) month, and follow-up visits at three (3) months, six (6) months and 12 months following EOT.
  Interventions: Combination Product: ST266 via Intranasal Delivery
- Cohort Two (Experimental): Three (3) subjects, ST266 400 µL administered by trans-cribriform intranasal device bilaterally (200 µL/nostril) once a day for 14 days with a follow-up visit at seven (7) days following EOT, a follow-up call at one (1) month, and follow-up visits at three (3) months, six (6) months and 12 months following EOT.
  Interventions: Combination Product: ST266 via Intranasal Delivery
- Cohort Three (Experimental): Three (3) subjects, 400 µL ST266 administered by trans-cribriform intranasal device bilaterally (200 µL/nostril) once a day for 28 days with a follow-up visit at seven (7) days following EOT, a follow-up call at one (1) month, and follow-up visits at three (3) months, six (6) months and 12 months following EOT.
  Interventions: Combination Product: ST266 via Intranasal Delivery

INTERVENTIONS:
Combination Product: ST266 via Intranasal Delivery — ST266 administered by non-invasive trans-cribriform intranasal delivery using the SipNose intranasal device.

SUMMARY:
The primary objective of this trial is to assess the safety of ST266 given by non-invasive intranasal trans-cribriform delivery to glaucoma suspect subjects with ocular hypertension, optic nerve cupping, or family history of glaucoma.

DETAILED DESCRIPTION:
This clinical trial is a dose escalating design in three (3) cohorts. In the first cohort, subjects will be treated with ST266 delivered using a non-invasive trans-cribriform intranasal delivery device daily for 14 days, in alternating single nostrils. If there are no SAEs and no pattern of concern in the AE's, the Investigator may proceed to the second cohort. In Cohort Two, subjects will be administered ST266 to each nostril daily for 14 days. As with the first cohort, if there are no safety concerns, the investigator may move on to the third cohort. In Cohort Three, subjects will be administered ST266 to each nostril daily for 28 days. All subjects will be followed for 12 months after the last dose of study drug. ST266 will be administered by a health care professional trained to deliver ST266 intranasally. No efficacy data will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form and HIPAA (Health Insurance Portability and Accountability Act) document.
2. Male or Female, Ages 20-75 years.
3. Must be clinically followed as a glaucoma suspect without evidence of glaucomatous damage.
4. Must have one of the following: 1) IOP ≤ 28 mmHg and at least one (1) IOP measurement > 21 mmHg, or 2) physiologic cupping of the optic nerve, or 3) a family history of glaucoma.
5. Two (2) normal visual fields (VF) both Swedish Interactive Threshold Algorithm - Short-wavelength Automated Perimetry (SITA-SWAP) and 24-2 VF prior to subject enrollment at the Baseline Visit.
6. Two (2) normal Ocular Coherence Tomography (OCT) (of macula and nerve fiber layer) prior to subject enrollment at the Baseline Visit.
7. Gonioscopy open to at least scleral spur with normal iris configuration.
8. Normal baseline neuro-cognitive testing.
9. Normal baseline Magnetic Resonance Imaging (MRI), including expected age-related changes, performed with and without contrast.
10. Cohort Three group only: Baseline Lumbar Puncture within normal limits.

Exclusion Criteria:

1. Females of Child Bearing Potential (FOCBP) who are pregnant or lactating or who will not abstain from sexual activity for 14 days prior to Visit 1, and willing to remain so through 30 days following completion of the subject's first menstrual cycle following the End of Treatment (EOT) Visit. Alternatively, a WOCBP who will not remain abstinent must have been using one of the following acceptable methods of birth control for the times specified:

   * IUD in place for at least three (3) months prior to Visit 1 until completion of the subject's first menstrual cycle following the EOT Visit.
   * Barrier method (condom or diaphragm) with spermicide for at least three (3) months prior to Visit 1 through completion of the subject's first menstrual cycle following the EOT Visit.
   * Stable hormonal contraceptive for at least three (3) months prior to Visit 1 through completion of the subject's first menstrual cycle following the EOT Visit. NOTE: For Depo-Provera injection contraceptives, the statement regarding first menstrual cycle following administration of the study product is not applicable as females receiving this form of contraception will not have menses.
   * In a monogamous relationship with a surgically sterilized (i.e., vasectomized) partner at least six (6) months prior to Visit 1.
   * Have undergone one of the following sterilization procedures at least six (6) months prior to Visit 1: Bilateral tubal ligation, Hysterectomy, Hysterectomy with unilateral or bilateral oophorectomy, Bilateral oophorectomy.
2. Unwillingness to submit a urine pregnancy test at screening if of childbearing potential.
3. Male subjects who refuse to use one of the following birth control methods:

   * Abstinence from the time of consent and through the duration of their participation in the protocol
   * Barrier method (condom or diaphragm) with spermicide from time of consent through the duration of their participation in the protocol
   * Surgical sterilization (vasectomy) at least 6 months prior to consent.
4. IOP greater than 29 mmHg in either eye.
5. Patients with high risk factors of ocular hypertension, such as thin central corneas, as identified by the Principal Investigator who may benefit from earlier treatment will be excluded.
6. Evidence of Angle closure.
7. Recent laser or incisional glaucoma surgery.
8. Subjects who are currently taking glaucoma medications. Subject who can safely stop taking these medications during washout period (4-6 weeks) may be considered.
9. Intranasal polyp or any head and/or neck neoplasm.
10. History of or evidence on physical examination including endoscopy of sinus or nasal pathology, nasal passage obstruction, chronic sinus infections, or severe seasonal allergies.
11. Currently using medications given intranasally.
12. Subject is taking any anticoagulant medication such as heparin, low molecular weight heparin, Coumadin, or antiplatelet agents including low dose aspirin.
13. History of stroke or Trans-Ischemic Attack (TIA) within the past five (5) years.
14. Neuro-cognitively impaired as assessed by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
15. Subjects who have participated in an investigational product trial within the past 30 days.
16. Subjects who refuse any part of the protocol assessments.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 18 months (entire duration of study)
  Safety will be determined by comparing the results of the screening tests at baseline and again at the end of the treatment period through the end of study. Adverse events (AEs) and Serious Adverse Events (SAEs) will be recorded. The primary safety variable is the incidence of subjects with any adverse event during the entire study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No